CLINICAL TRIAL: NCT06444087
Title: Patient's Perspective on the Evolution of Hidradenitis Suppurativa Burden After Secukinumab Initiation: a French Multicentric Prospective Observational Study
Brief Title: Patient's Perspective on the Evolution of Hidradenitis Suppurativa Burden After Secukinumab Initiation
Acronym: SPECTRA
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457MFR01
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: secukinumab; Hidradenitis Suppurativa; HS; NIS; France
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- secukinumab: Patients prescribed with secukinumab
  Interventions: Other: secukinumab

INTERVENTIONS:
Other: secukinumab — This is an observational study. There is no treatment allocation. The decision to initiate secukinumab will be based solely on clinical judgement.

SUMMARY:
The primary objective of this non-interventional study is to describe the evolution of Hidradenitis suppurativa (HS) symptoms 12 months after secukinumab initiation based on the patients' assessment of pain, oozing, and bad smell.

DETAILED DESCRIPTION:
This study is a prospective (primary data), national, descriptive, non-interventional, multicentre study conducted by medical practice and hospital-based dermatologists across different geographical regions in France.

This real-world study does not change the physician-patient relationship or patient management or follow-up. Physicians remain free with their prescriptions and patient follow-up procedures. In fact, secukinumab initiation and all treatment decisions will be made according to routine medical care and independently of study participation.

Recruited patients will be longitudinally followed-up for the duration of the study, up to 24 months (± 3 months) after secukinumab initiation or secukinumab treatment discontinuation before the end of the 24 months of follow-up (early discontinuation).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 18 years old,
2. Patients who do not object to participation in the study,
3. Diagnosis of HS clinically confirmed,
4. Initiation of secukinumab treatment for HS in compliance with the summary of product characteristics,
5. The physician's decision to initiate secukinumab has been taken according to his/her own practice and regardless of study participation.

Exclusion Criteria:

1. Patients with any medical or psychological condition which, in the physician's opinion, may prevent participation in the study,
2. Patients participating in a clinical trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include male and female patients (aged ≥ 18 years) with a diagnosis of HS and for whom the decision to initiate treatment with secukinumab was made independently of the study.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving at least 30% reduction of the NRS score for at least one the assessed symptoms | Baseline, month 12
  Patients will provide an assessment of pain, oozing and bad smell based on three numeric rating scales (NRS). The most common form of the scale is a horizontal line with a numeric scale ranging from 0 to 10, 0 corresponding to "no symptoms" and 10 being the worst possible symptom. At each visit, these three assessments will cover the last seven days.

SECONDARY OUTCOMES:
Proportion of patients achieving at least a 30% reduction of NRS | Baseline, month 3, month 6, month 18 and month 24
  Proportion of patients achieving at least a 30% reduction of NRS for at least one of the evaluated symptoms (pain, oozing and bad smell) and the proportion of patients achieving at least a 30% reduction of NRS for each symptom evaluated separately (pain, oozing and bad smell)
Proportion of patients achieving at least a 5-point reduction of the Dermatology Life Quality Index (DLQI) | Baseline, month 3, month 6, month 18 and month 24
  The DLQI consists of ten questions regarding patients' perception of the impact of their disease on different aspects of their health-related quality of life (symptoms and feelings, impact on daily activities, leisure, work, school, personal relationships, and problems with treatment) over the last seven days. The highest possible total score for the DLQI is 30 and higher scores indicate a more severe impact on quality of life.
Proportion of patients maintaining the improvement up to 24 months of the response of the Impact of Hidradenitis Suppurativa on daily life compared to baseline | Baseline, up to 24 months
  The impact of Hidradenitis Suppurativa (HS) on daily life will be studied using seven additional questions on the symptoms experienced by the patient and the impact of HS on daily life over the past three months: physical and psychological fatigue, anxiety, sleep quality, discomfort with dressing, discomfort with washing, and sex and love life. Responses will be collected at each visit by a four-point Likert scale. The improvement will be defined by the decrease of at least one point on the Likert scale between the enrolment visit and the follow-up visits.
Proportion of patients having stopped at tobacco, alcohol and cannabis use | Baseline, month 3, month 6, month 18 and month 24
  The proportion of patients having stopped at least one of these substances during follow-up will be calculated, and as well as the proportion of patients having stopped one of these substances without using them again until the end of follow-up.
Absenteeism due to Hidradenitis Suppurativa | Baseline, month 3, month 6, month 18 and month 24
  Absenteeism due to HS will be measured by the number of days off taken and the number of days on sick leave over the last three months (enrolment visit and visit at 3 months) or since the last visit (visits at 6, 12, 18 and 24 months). The number of days and its evolution since enrolment will be presented at each visit.
Proportion of patients achieving at least a 5-point reduction of FDLQI compared to the baseline | Baseline, month 3, month 6, month 18 and month 24
  The family member's quality of life will be measured using the FDLQI. The FDLQI is a 10-item-questionnaire with a total score resulting in a maximum of 30 and a minimum of 0 (the higher the score, the more quality of life is impaired). The questionnaire will be proposed to one of the family members (one per patient, the same person throughout the study) going with the patient to the baseline visit and 3, 6, 12, 18 and 24 months after secukinumab initiation. The assessment will refer to the last seven days.
Secukinumab dose regimen prescribed at baseline | Baseline
  Secukinumab dose regimen prescribed at baseline to describe the use of secukinumab.
Proportion of patients receiving up-titration or down-titration | Month 3, month 6, month 12, month 18 and month 24
  Proportion of patients receiving up-titration (q4w-to-q2w) or down-titration (q2w-to-q4w) and proportion of patients receiving more than one up-and/or down-titration
Time spent under each treatment regimen | Up to 24 months
  Time spent under each treatment regimen (q4w and q2w) and reason for change
Total duration of secukinumab treatment | Up to 24 months
  Total duration of secukinumab treatment (i.e. time elapsed until treatment is discontinued), reason for discontinuation
Proportion of patients with at least one temporary discontinuation | Up to 24 months
  Proportion of patients with at least one temporary discontinuation and its reason
Proportion of patients taking all prescribed doses | Up to 24 months
  Proportion of patients taking all prescribed doses to measure the treatment compliance
Proportion of patients achieving a reduction in IHS4 | Baseline, month 3, month 6, month 12, month 18 and month 24
  Proportion of patients achieving at least 55%, 75% and 100% reduction in International Hidradenitis Suppurativa Severity Score System (IHS4) (IHS4-55, 75, 100).
  The IHS4 score corresponds to: (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of drainage tunnels (fistulas/sinuses) multiplied by 4]. A score of 3 or less corresponds to mild HS, a score of 4 to 10 to moderate HS and a score of 11 or more to severe HS
Evolution of AN count | Baseline, month 3, month 6, month 12, month 18 and month 24
  Evolution of AN count (total abscesses and inflammatory nodules)
Percentages of patients with onset or worsening of flares | Baseline, month 3, month 6, month 18 and month 24
  Percentages of patients with onset or worsening of flares will be described from the data concerning flares collected by the physician at each visit.
Proportion of patients who achieved at least a 30% reduction in the NRS score (pruritus) | Baseline, month 3, month 6, month 18 and month 24
  Itching due to pruritus will be evaluated using an 11-point NRS scale with 0 being "no itch" and 10 being the worst itch imaginable.
Proportion of patients receiving at least one medication for HS | Month 3, month 6, month 18 and month 24
  Treatments of interest will include systemic antibiotics, pain medications and psychotropic drugs.
Proportion of patients who had a surgical procedure | Up to 24 months
  Proportion of patients who had a surgical procedure will be provided
Proportion of patients with stable/increased/decreased dressing used since the baseline visit | Baseline, month 3, month 6, month 18 and month 24
  Use of dressings and protections for wound care after secukinumab initiation, evaluated by the use of dressings and protections in the seven days prior to visits (data collected by the patient)
Number of patients by reasons for secukinumab initiation | Baseline
  Description of the reasons for secukinumab initiation (e.g.: patient complaints, clinical symptoms, safety events) declared by the participating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- France (22):
  - Novartis Investigative Site, Nice, France
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Calais
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lorient
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rodez
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Mandé
  - Novartis Investigative Site, Saint-Pierre
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vannes

IPD SHARING:
Plan to Share IPD: No